CLINICAL TRIAL: NCT05277376
Title: Ultraviolet Filter Bemotrizinol (BEMT): Clinical Pharmacokinetics Evaluation in a Topical Maximum Usage Trial (MUsT)
Brief Title: Pharmacokinetic (PK) Evaluation of Bemotrizinol (6%) in a Sunscreen Maximum Usage Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: BEMT-001 (Part 2)
Record Dates: First submitted 2022-02-11; First posted 2022-03-14 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-03

CONDITIONS: Pharmacokinetics; Absorption; Chemicals
Keywords: Sunscreen Maximum Usage Trial; MUsT
MeSH Terms: interventions — bis-ethylhexyloxyphenol methoxyphenyl triazine

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, 3-arm study in 162 healthy adult subjects with the following objective: Primary: To assess the systemic absorption and pharmacokinetics of BEMT from 3 different market image sunscreen drug formulations containing 6% BEMT under maximal-use conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BEMT Formulation SU-E-101413-85 (Active Comparator): PK evaluation of 6% BEMT after multiple applications of a topical sunscreen formulation.
  Interventions: Drug: Bemotrizinol (6%)
- BEMT Formulation SU-E-101413-87 (Active Comparator): PK evaluation of 6% BEMT after multiple applications of a topical sunscreen formulation.
  Interventions: Drug: Bemotrizinol (6%)
- BEMT Formulation SU-E-101413-89 (Active Comparator): PK evaluation of 6% BEMT after multiple applications of a topical sunscreen formulation.
  Interventions: Drug: Bemotrizinol (6%)

INTERVENTIONS:
Drug: Bemotrizinol (6%) — Active sunscreen ingredient (Broad spectrum UV-Filter)
  Other Names: PARSOL SHIELD; BEMT; bis-ethylhexyloxyphenol methoxyphenyl triazine

SUMMARY:
An open-label, randomized, 3-arm study in 162 healthy adult subjects with the following primary objective: To assess the systemic absorption and pharmacokinetics of BEMT from 3 market image sunscreen formulations under maximal-use conditions.

DETAILED DESCRIPTION:
This study is an open-label, randomized, 3-arm pivotal study to evaluate the pharmacokinetics of BEMT after multiple applications of a topical sunscreen formulation in healthy adult subjects.162 subjects will be enrolled (54 subjects per study drug formulation arm) in order to achieve a minimum of 150 completers (50 completers in each arm).There will be an adequate representation of male and female subjects, subjects of all ages (including a sufficient number of elderly subjects), and subjects of different races.

All 162 subjects will randomized at Day -1 and assigned to a treatment arm before study drug application on Day 1.

Treatment: Approximately 2 mg of a sunscreen formulation (approximately 0.12 mg BEMT) per 1 cm2 of body surface area will be applied topically 4 times per study day for 4 days (every 2 hours for 6 hours) to at least 75% of the body surface area.

Subjects will be randomly assigned to 1 of 3 treatment groups within each subgroup; Thus each subject will receive 1 of the sunscreen formulations. Treatment groups:

Treatment Group B: 54 subjects; Treatment: BEMT, PARSOL Shield, 6%, with suitable solubilizers; SU-E-101413-85: Sunscreen oil formulation with 10% ethanol Treatment Group C: 54 subjects; Treatment: BEMT, PARSOL Shield, 6%, with suitable solubilizers, SU-E-101413-87: oil-in-water (O/W) formulation Treatment Croup D: 54 subjects: Treatment: BEMT, PARSOL Shield, 6%, with suitable solubilizers, SU-E-101413-89: water-in-oil (W/O) formulation

Dosing will between 07:00 and 10:00 hours followed by 3 more applications at 2, 4, and 6 hours after the 1st application each day. Blood samples collected from before the 1st application through 96 hours after the 1st application.

The following noncompartmental PK parameters will be calculated for each subject using the plasma BEMT concentration-time data (data permitting):

* Cmax: Maximum observed concentration; computed for Overall, Day 1, and Day 4
* Tmax: Time of Cmax; computed for Overall, Day 1, and Day 4
* C2h: The concentration at 2 hours after the 4th daily study drug application; computed for Days 1, 2, 3, and 4
* Ctrough: The concentration at the end of the study day; computed for Days 1, 2, 3, and 4 at 23.5, 47.5, 71.5, and 96 hours, respectively
* AUC: Area under the concentration-time curve from before the first daily dose to the last measurable concentration in the time interval; computed for Overall, Day 1, and Day 4
* λz: Apparent elimination rate constant, computed from all relevant concentration data following the last study drug application on Day 4
* t1/2: Terminal elimination half-life, computed from λz

With the time intervals for Overall and Days 1, 2, 3, and 4 defined as:

* Overall = 0 to 264 hours
* Day 1 = 0 to 23.5 hours
* Day 2 = 23.5 to 47.5 hours
* Day 3 = 47.5 to 71.5 hours
* Day 4 = 71.5 to 96 hours

Note: If all concentrations for a subject are below the limit of quantitation (BLQ), then only the C2h and Ctrough parameters will be reported for that subject.

.

ELIGIBILITY:
Inclusion Criteria:

1. Subject signs an IRB-approved written informed consent form (ICF) and privacy language as per national regulations (e.g., Health Insurance Portability and Accountability Act [HIPAA] authorization) before any study-related procedures are performed.
2. Subject is a healthy man or woman, ≥18 years of age and who has a body mass index of 18.5 to 29.9 kg/m2, inclusive, at Screening.
3. Subject has normal medical history findings, clinical laboratory results, vital sign measurements, 12-lead electrocardiogram (ECG) results, and physical examination findings at Screening or, if abnormal, the abnormality is not considered clinically significant (as determined and documented by the investigator or designee).
4. Subject has a negative test result for alcohol and drugs of abuse at Screening and Check-in (Day -1).
5. Female subject is surgically sterile (hysterectomy, bilateral salpingo-oophorectomy, bilateral tubal ligation) or has a negative serum pregnancy test result before entry into the study and practices an adequate method of birth control (e.g., oral or parenteral contraceptives, hormonal or nonhormonal intrauterine device, barrier, abstinence) during the study and until 90 days after the last application of study drug.
6. Male subject agrees to refrain from sexual activity with female partners unless an acceptable method of birth control is used by both partners. Male subject is surgically sterile or agrees to use barrier contraception (condom with spermicide), and refrain from sperm donation, from the first application of study drug until 90 days after the last application of study drug.
7. Subject has a negative SARS-CoV-2 test result at Check-in (Day -1).
8. Subject is highly likely (as determined by the investigator) to comply with the protocol-defined procedures and to complete the study.

Exclusion Criteria:

1. Subject who participated in Part 1 of the present maximum usage trial (MUsT).
2. Subject has broken, irritated, or unhealed skin.
3. Subject has an active sunburn.
4. Subject has used a tanning bed in the previous 4 weeks.
5. Subject has known skin or autoimmune disease(s).
6. Subject is anemic or has any chronic condition(s) that may impact blood sample collection.
7. Women who are pregnant, breastfeeding, or planning to become pregnant during the study or during the 30 days after study drug administration. All female subjects will undergo a serum pregnancy test at Screening, on Day -1, and before discharge from the CRU.
8. Subject has any underlying disease or surgical or medical condition (e.g., cancer, HIV, severe hepatic or renal impairment) that could put the subject at risk or would normally prevent participation in a clinical study.
9. Subject has known or suspected allergies or sensitivities to any components of the sunscreen formulation.
10. Subject has clinical laboratory test results (hematology and serum chemistry) at Screening that are outside the reference ranges provided by the clinical laboratory and considered clinically significant by the investigator.
11. Subject has used alcohol-, caffeine-, or xanthine-containing products, Seville oranges (sour), grapefruit, or grapefruit juice, within 72 hours before first study drug application.
12. Subject has a positive test result at Screening for HIV type 1 or 2 antibody, hepatitis C virus antibodies, or hepatitis B surface antigen.
13. Subject is unable or unwilling to undergo multiple venipunctures for blood sample collection because of poor tolerability or poor venous access.
14. Subject has used any product(s) containing bis-ethylhexyloxyphenol methoxyphenyl triazine (BEMT), such as sunscreen products, hand or body moisturizing lotion, makeup or foundation, hair care product, lip balm, or lipstick within 14 days before Check-in (Day -1) and at any time before End-of-Study procedures.
15. Subject is unable or unwilling to tolerate the scent of sunscreen and the body coverage with sunscreen (i.e., oily appearance and sensation of sunscreen) for the duration of the treatment period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female, male
Enrollment: 162 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of BEMT | 4 days
  Assess Cmax (maximum observed drug concentration) of BEMT in plasma from three high-penetrating sunscreen formulations under maximal-use conditions computed for Overall, Day 1, and Day 4. With the time intervals for Overall and Days 1, 2, 3, and 4 defined as: Overall = 0 to 264 hours; Day 1 = 0 to 23.5 hours; Day 2 = 23.5 to 47.5 hours; Day 3 = 47.5 to 71.5 hours; and Day 4 = 71.5 to 96 hours.
Time of Maximum Observed Concentration (Tmax) of BEMT | 4 days
  Assess the time at which the maximum concentration (Cmax) of BEMT occurs in plasma from three high-penetrating sunscreen formulations under maximal-use conditions; Overall, Day 1, and Day 4. With the time intervals for Overall and Days 1, 2, 3, and 4 defined as: Overall = 0 to 264 hours; Day 1 = 0 to 23.5 hours; Day 2 = 23.5 to 47.5 hours; Day 3 = 47.5 to 71.5 hours; and Day 4 = 71.5 to 96 hours.
Concentration of BEMT at 2 hours (C2h) after the 4th daily study drug application | 4 days
  Assess the plasma concentration of BEMT at 2 hours after the 4th daily study drug application; computed for Days 1, 2, 3, and 4
Concentration at the end of the study day (Ctrough) | 4 days
  Assess plasma concentration of BEMT at the end of the study day, computed for Days 1, 2, 3, and 4 at 23.5, 47.5, 71.5, and 96 hours, respectively
Area under the concentration-time curve (AUC) | 4 days
  Assess area under the concentration-time curve from before the first daily dose to the last measurable concentration in the time interval); computed for Overall, Day 1, and Day 4.
Apparent elimination rate constant (λz) | 4 days
  Assess the apparent elimination rate constant for BEMT in plasma; computed from all relevant concentration data following the last study drug application on Day 4.
Terminal elimination half-life (t1/2) | 4 days
  Assess the time required for BEMT to decrease by a factor of one-half in plasma computed from λz, which will be computed from all relevant concentration data following the last study drug application on Day 4.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Boston, MSN, APNP, Principal Investigator — Spaulding Clinical Research LLC
Locations (1):
- Spaulding Clinical Research LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No